CLINICAL TRIAL: NCT06262893
Title: Effect of Dexamethasone Adjuvant in Combined Supraclavicular Block and Suprascapular Block Versus Interscalene Block in Patients Undergoing Shoulder Arthroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shoulder nerve blocks
Record Dates: First submitted 2023-12-26; First posted 2024-02-16 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Arthroscopy Blocks; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene block in shoulder arthroscopy (Active Comparator)
  Interventions: Procedure: Shoulder arthroscopy blocks
- Combined Supraclavicular block and suprascapular block in shoulder arthroscopy (Active Comparator)
  Interventions: Procedure: Shoulder arthroscopy blocks

INTERVENTIONS:
Procedure: Shoulder arthroscopy blocks — Effect of dexamethasone adjuvant in combined supraclavicular block and suprascapular block versus Interscalene block in patients undergoing shoulder arthroscopy.

SUMMARY:
In this study the investigators aim to compare the effect of the suprascapular- supraclavicular nerve block in association with dexamethasone to that of the interscalene brachial plexus block on analgesic effect during arthroscopic shoulder surgery, as postoperative pain scores ,postoperative consumption of analgesic rescue medications and diaphragmatic excursion assessment.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1,2.

  * Age 18 years or older
  * Elective shoulder arthroscopic surgery under general anesthesia and nerve block performed preoperatively.

Exclusion Criteria:

* • Patient refusal

  * Serious cardiac arrhythmias (including atrial fibrillation) or unstable coronary artery disease.
  * Use of drugs that act on the autonomic nervous system (including β- blockers).
  * Coagulation disorders..
  * Anatomical disorders and/or neuropathic disease.
  * BMI above 40.
  * History of substance abuse.
  * Chronic use of psychotropic and/or opioid.
  * History of psychiatric diseases needing treatment.
  * Allergy to any drug in the study protocol.
  * Failure of nerve block performed in the preoperative block room when tested prior to entering the operating room (i.e. lack of loss of sensation to ice at the shoulder incision level).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia by visual analog scale (VAS). | 48 hours
  The
  primary outcome of this study will be to evaluate and compare between suprascapular-supraclavicular nerve block in association with dexamethasone to that of the interscalene brachial plexus block on postoperative analgesia by vas score during 48h postoperatively ( 2h , 6h , 12h, 24h and 48h).
  The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Diaphragmatic excursion | 1hour postoperatively
  Assessment of diaphragmatic excursion by ultrasound preoperatively and 1hour postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No